CLINICAL TRIAL: NCT00798551
Title: Emergency Department Interventions to Improve Blood Pressure Follow-up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0519-07-EP
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risk counseling (Other): Risk counseling regarding elevated blood pressure
  Interventions: Behavioral: Risk counseling

INTERVENTIONS:
Behavioral: Risk counseling — cardiovascular risk counseling regarding elevated blood pressure

SUMMARY:
Hypertension affects approximately 65 million people in the United States and approximately 20 million individuals remain undiagnosed. In Emergency Room visits, many as one third of the patients were noted to have elevated BP readings, two thirds of which could benefit from further therapy or closer clinic follow-up. However primary care follow-up after discharge with an elevated BP is surprisingly low. The purpose of this study is to measure the follow-up rate after the Emergency Room visit in individuals identified with elevated blood pressure after a brief counseling regarding risks of elevated blood pressure.

DETAILED DESCRIPTION:
Hypertension is a very common disease, affecting approximately 65 million people in the United States. As many as 30 % of people with hypertension, approximately 20 million individuals, remain undiagnosed. As many as one third of patients seen in ED were noted to have elevated BP readings in prior studies. Approximately 5% of emergency department (ED) patients have severely elevated blood pressure. Prior studies suggest that as many as two thirds of ED patients with elevated BP can benefit from further therapy or closer clinic follow-up. However primary care follow-up after ED discharge with an elevated BP is surprisingly low. The purpose of this study is to measure the follow-up rate after the ED visit in individuals identified with elevated blood pressure after a brief counseling regarding risks of elevated blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* diastolic BP 90 mm Hg or systolic BP 140 mm Hg
* diabetes and chronic kidney disease who have a diastolic BP 80 mm Hg or systolic BP 130 mm Hg

Exclusion Criteria:

* unable/unwilling to provide informed consent
* acute anxiety state
* Any subject on pain medication which compromises their ability to consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04-16 (Actual); Primary Completion 2010-12-20 (Actual); Study Completion 2010-12-20 (Actual)

PRIMARY OUTCOMES:
Follow-up with Primary care physician | one month
  The purpose of this study is to measure the follow-up rate after the ED visit in individuals identified with elevated blood pressure after a brief counseling regarding risks of elevated blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Srikar R Adhikari, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Result] Backer HD, Decker L, Ackerson L. Reproducibility of increased blood pressure during an emergency department or urgent care visit. Ann Emerg Med. 2003 Apr;41(4):507-12. doi: 10.1067/mem.2003.151. PMID 12658251
- [Result] Karras DJ, Ufberg JW, Heilpern KL, Cienki JJ, Chiang WK, Wald MM, Harrigan RA, Wald DA, Shayne P, Gaughan J, Kruus LK. Elevated blood pressure in urban emergency department patients. Acad Emerg Med. 2005 Sep;12(9):835-43. doi: 10.1197/j.aem.2005.04.015. PMID 16141017
- [Result] Preston RA, Baltodano NM, Cienki J, Materson BJ. Clinical presentation and management of patients with uncontrolled, severe hypertension: results from a public teaching hospital. J Hum Hypertens. 1999 Apr;13(4):249-55. doi: 10.1038/sj.jhh.1000796. PMID 10333343